CLINICAL TRIAL: NCT06154486
Title: Evaluation of Gastric Content of Volunteers Fasting and Using Semaglutide: an Observational and Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: 69273023.7.0000.0071
Record Dates: First submitted 2023-09-14; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-09

CONDITIONS: Pneumonia, Aspiration; Anesthesia
Keywords: gastric ultrasound; GLP-1 receptor agonists
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- semaglutide group: patients without risk factors for gastroparesis, fasting for at least 8 hours, BMI less than 30 and currently using semaglutide
  Interventions: Drug: semaglutide use
- control group: patients without risk factors for gastroparesis, fasting for at least 8 hours, BMI less than 30 and who have never used semaglutide or another GLP-1 analogue

INTERVENTIONS:
Drug: semaglutide use — patient using semaglutide for at least 7 days
  Other Names: control group
  Groups: semaglutide group

SUMMARY:
Medicines with peptide-1 receptor agonist action similar to glucagon (GLP-1) are a modern therapeutic option for obesity and diabetes mellitus. Semaglutide is a representative of this class medication whose mechanism of action can result in the slowing of gastric emptying and reduced gastric motility, a scenario that can increase the risk of pulmonary aspiration in individuals undergoing anesthesia and despite adequate fasting. Given the severity of the occurrence of bronchoaspiration, the action biological analysis of GLP-1 analogues on gastric function and incremental use of these medications, through gastric ultrasound, we will aim to evaluate the gastric contents of volunteers who do not have risk factors for bronchoaspiration, who will not undergo anesthesia, but are with the fasting recommended for this purpose and are using semaglutide, an analogue of GLP-1. Our hypothesis is that the majority of individuals using these medications have a full stomach even during fasting times recommended in the literature. In view of this, for this population we must adapt safety criteria during the anesthetic procedure.

DETAILED DESCRIPTION:
INTRODUCTION

Obesity and type 2 diabetes mellitus constitute a global public health problem. Medications with glucagon-like peptide-1(GLP-1) receptor agonist action are a modern therapeutic option for both diseases. Liraglutide, semaglutide and dulaglutide are some representatives of this drug class, whose mechanism of action results in slowing gastric emptying, reduced gastric motility, and increased gastric volume These effects are implicated in both weight loss and the occurrence of adverse events such as nausea, vomiting, acute gastroparesis and gastroesophageal reflux disease (GERD) The presence of gastric contents during the anesthetic procedure can lead to pulmonary aspiration and the development of chemical pneumonitis, a potentially fatal complication. To avoid this risk, in healthy patients, an 8-hour fast for solids and 2 hours for clear liquids. However, when there is a risk factor for slow gastric emptying, despite adequate fasting, the stomach may present residues and bedside ultrasound is an effective, non-invasive and quickly to measure this content and stratify the risk of aspiration Due to the lack of studies demonstrating that the use of GLP-1 analogue can increase the risk of aspiration in individuals who are fasting adequately to receive anesthesia, there is no formal recommendation for performing gastric ultrasound in the preoperative period, nor for the suspension of these medications. Some institutions empirically recommend suspension preoperatively.

Given the severity of the occurrence of bronchoaspiration, the biological action of GLP-1 analogues on gastric function and the incremental use of these medications, it is necessary to better understand the gastric contents of individuals fasting and using a GLP-1 analogue. GLP-1. Thus, through ultrasound, we will aim to evaluate the gastric contents of volunteers who do not have risk factors for bronchoaspiration, who will not undergo anesthesia, but are fasting recommended for this purpose and are using semaglutide, a GLP-1 analogue.

Our hypothesis is that the majority of individuals using these medications have a full stomach even with the fasting times recommended in the literature. In view of this, for this population we must adapt safety criteria during the anesthetic procedure.

Objectives Primary objective The primary objective is to evaluate the prevalence of a full stomach through gastric ultrasound examination in volunteers who use semaglutide and are fasting for at least 8 hours for solids and 2 hours for clear liquids. As a control group, we will use volunteers who do not use semaglutide.

Secondary objectives The secondary objectives consist of evaluating whether the demographic characteristics of the volunteers, the time of medication use, the time elapsed since the last dose of semaglutide received, the dose and regimen of medication use, the reason for using the medication, the presence Symptoms such as nausea, vomiting, loss of appetite and sensation of gastric fullness can influence gastric emptying when these individuals are evaluated by ultrasound.

Study Design Observational, cross-sectional, non-interventional study

study population

30 volunteers will be included in the study, of which 15 must be currently using semaglutide and 15 must not be using the medication. The gastric ultrasonography will be performed at Hospital Israelita Albert Einstein, in the radiologist medicine sector, by an anesthesiologist with experience in gastric ultrasonography. The images will be registered in the picture archiving and communication system and reviewed by a radiologist.

Sample size calculation Based on the literature, individuals in the control group presented an area of residual liquid in the stomach ranging from 3cm² to 7cm² with a median area of 5.1cm², which respectively provide 32.4ml, 90.8ml and 63.1ml of liquid volume. residual after 8 hours of fasting, assuming an average increase of at least 20ml of fluid in patients using semaglutide, with 95% confidence and 80% power, the sample required to carry out the study is 14 patients in each group. To compensate for any losses, we will increase the sample by 10%, leaving 15 volunteers in each group.

METHODS Study outcomes Primary outcome Compare the prevalence of a full stomach, after fasting for at least 8 hours for solids and 2 hours for clear liquids, through gastric ultrasound in volunteers using semaglutide with those who do not use the medication. The outcome will be binary: a full stomach includes the visualization of solids on gastric ultrasonography or a volume of clear liquids greater than 1.5ml/kg It will be considered an empty stomach when no content or clear liquids are visible inferior to 1.5ml/kg

Secondary outcomes

* Assess the demographic characteristics of the volunteers.
* Describe the dose and regimen of medication use.
* Describe the reason for using the medication.
* Describe the presence of symptoms such as nausea, vomiting and sensation of gastric fullness, loss of appetite, early satiety and abdominal pain.
* Describe the use of other medications.

Risk factors for bronchoaspiration

* Diabetes Mellitus with peripheral neuropathy or history of gastroparesis.
* Obesity. Defined as body mass index (BMI) inferior to 30 kg/m2.
* Active cancer.
* Gastroesophageal Reflux Disease.
* Use of opioids.
* History of surgery for obesity.
* Neurological disease.
* Chronic or acute kidney disease.
* Symptomatic hypothyroidism.

Technical limitation for evaluation of gastric contents by ultrasonography

* Previous gastric surgery such as partial gastrectomy or gastric bypass.
* Massive hiatus hernia.

Proper fasting

Fasting will be considered adequate:

* general diet: 8 hours
* Clear liquids (water, juices without lumps): 2 hours

Types of GLP-1 analogue

The following drugs will be considered:

• Semaglutide: Ozempic®️, Wegovy®️

Protocol for performing gastric ultrasonography

It consists of scanning the abdomen in the sagittal plane in the dorsal decubitus position at 45 degrees in the supine position and in the right lateral decubitus position with a curvilinear, low-frequency ultrasound probe(2 to 5 mHz) and locating the gastric antrum, through the identification of the main points of reference - left lobe of the liver and a main vessel, aorta or inferior vena cava. Gastric emptying will be assessed quantitatively and qualitatively, through assessment of the composition of its contents and measurement of gastric volume, respectively.

The qualitative assessment will assess whether the stomach is empty, with clear liquid or with solids. The stomach is considered empty when the antrum presents itself with the anterior and posterior walls juxtaposed, denoting a "buffalo eye" or "target" pattern, a characteristic attributed by the identification of a hypoechoic, thick external ring. The antrum may appear empty in the supine position and fluid-filled in the right lateral decubitus position. The volume of liquid must be measured in this position and if it is less than 1.5 ml/kg (average of 100ml in adults) it is considered normal in fasting individuals and the risk of bronchoaspiration is considered low. On the other hand, the visualization of liquid both in the supine position and in the right lateral decubitus position is suggestive of a large gastric volume. When the liquid measurement is greater than 1.5 ml/kg, the patient is at high risk for bronchoaspiration.

Whenever clear liquids are visualized, gastric volume is measured using the cross-sectional area of the gastric antrum(AA) using the external wall of the stomach, which has a linear correlation with gastric volume. This is performed in the right lateral decubitus position with two perpendicular diameters of the antrum, from serosa to serosa, the longitudinal or craniocaudal diameter(CC) and the anteroposterior diameter (AP) or using the ellipse formula developed by Bolondi where AA=(CC× AP × π) /4. With the value of π = 3.14. After calculating the AA, the total stomach volume ("predicted volume") will be evaluated in each volunteer with a previously tested and validated mathematical model, in which the stomach volume(ml) = 27 + 14.6 x AA (cm2) - 1.28 age (in years).

Collected variables Demographic data will be collected. Ultrasound images will be registered in the radiology picture archiving and communication system. Data will be collected in printed clinical records and/or an electronic form specifically developed for the study, using the REDCap@ (Research Electronic Data Capture) electronic form. The authors will be responsible for monitoring the data.

Demographic and baseline data.

* Verification of inclusion and exclusion criteria.
* Applicability and date of application of the informed consent form
* Date of birth.
* Age (in years).
* Gender.
* Ethnicity.
* Weight (in kg).
* Height (in cm).
* BMI (in kg/m2).
* Date of inclusion in the study.

Data regarding the GLP-1 analogue

* Semaglutide
* Ozempic®️
* Wegovy®️
* Administration dosage:
* Time of medication use in months or weeks, when time of use is less than 1 month.
* Previous use of semaglutide?
* Previous use of another medication from the GLP-1 analogue class?
* Reason for using the medication:

Clinical symptoms of gastroparesis

* Nausea
* Vomiting
* Abdominal pain
* Sensation of gastric fullness
* Early satiety
* Loss of appetite

Use of other medications

Data regarding gastric ultrasound examination

• Qualitative check

* Full stomach - solid residue or clear liquid volume> 1.5 ml/kg
* Empty stomach - no content or volume of clear liquid Volume ≤ 1.5 ml/kg

STATISTICAL ANALYSIS Included patients will be divided into two groups according to the use or not of Semaglutide and the gastric residue found: a full stomach or an empty stomach. Differences between groups in relation to continuous numerical variables will be analyzed using the Student t test (normal distribution) or Mann-Whitney U test (variables not normally distributed). Proportions will be compared using the Chi-square test or Fisher's Exact Test, All significance probabilities (p values) presented will be two-tailed. p-values will be considered statistically significant when less than 0.05. All analyzes will be performed using the software R 3.4.1 (R Foundation for Statistical Computing, Vienna, Austria)

SAFETY AND ETHICAL CONSIDERATIONS Risks and benefits Abdominal ultrasound is a non-invasive exam that does not emit radiation. There is no evidence to support that the use of ultrasound can cause any harm to health. The research participant may experience some discomfort related to fasting for 8 hours for solids and 2 hours for liquids.

There are risks related to the loss of data confidentiality and the research team is responsible for taking all precautions to ensure data confidentiality.

This study may benefit individuals who use this medication when undergoing anesthesia. According to the results of this study, suspension of this medication preoperatively or other safety measures may be recommended.

Approval from ethical and regulatory authorities The study was approved by the Institutional review Board (IRB) and written consent from the patient will be requested.

Data confidentiality The patient will be identified by the corresponding number on the electronic data collection form. The data obtained must be kept confidential by the researchers and will be stored on the REDCAP Platform, which allows restricted access to information, according to security levels and individualized logins.

ELIGIBILITY:
Inclusion Criteria:

* • Adult individuals (aged 18 or over).

  * Individuals currently using semaglutide.
  * Individuals fasting for at least 8 hours for solids and 2 hours for clear liquids without residue.

Exclusion Criteria:

* Pregnant women and postpartum women.

  * Individuals with technical limitations to perform gastric content assessment using ultrasonography
  * Presence of risk factors for gastroparesis.
  * Use of drugs from the prokinetic class, which accelerate gastric emptying, such as bromopride, metoclopramide and domperidone.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 30 volunteers will be included in the study, of which 15 must be currently using semaglutide and 15 must not be using the medication. The gastric ultrasonography will be performed at Hospital Israelita Albert Einstein, in the radiologist medicine sector, by an anesthesiologist with experience in gastric ultrasonography. The images will be registered in the picture archiving and communication system and reviewed by a radiologist.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
prevalence of full stomach after fasting for at least 8 hours | 1 day
  Compare the prevalence of a full stomach, after fasting for at least 8 hours for solids and 2 hours for clear liquids, through gastric ultrasound in volunteers using semaglutide with those who do not use the medication. The outcome will be binary: a full stomach includes the visualization of solids on gastric ultrasonography or a volume of clear liquids greater than 1.5ml/kg.
  It will be considered an empty stomach when no content or clear liquids are visible inferior to 1.5ml/kg.

SECONDARY OUTCOMES:
demographic distribution | 1 day
  • Assess the demographic characteristics
medication information | 1 day
  Describe the dose and regimen of medication use and reason for using the medication.
Incidence of symptoms associated with medication use | 1 day
  Describe the presence of symptoms such as nausea, vomiting and sensation of gastric fullness, loss of appetite, early satiety and abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: veronica fialho, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalra S, Bhattacharya S, Kapoor N. Contemporary Classification of Glucagon-Like Peptide 1 Receptor Agonists (GLP1RAs). Diabetes Ther. 2021 Aug;12(8):2133-2147. doi: 10.1007/s13300-021-01113-y. Epub 2021 Jul 15. PMID 34268675
- [Background] Halawi H, Khemani D, Eckert D, O'Neill J, Kadouh H, Grothe K, Clark MM, Burton DD, Vella A, Acosta A, Zinsmeister AR, Camilleri M. Effects of liraglutide on weight, satiation, and gastric functions in obesity: a randomised, placebo-controlled pilot trial. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):890-899. doi: 10.1016/S2468-1253(17)30285-6. Epub 2017 Sep 27. PMID 28958851
- [Background] Almustanyir S, Alhabeeb H, AlHusseini N, Al Thow M. Gastroparesis With the Initiation of Liraglutide: A Case Report. Cureus. 2020 Nov 28;12(11):e11735. doi: 10.7759/cureus.11735. PMID 33403167
- [Background] Warner MA, Meyerhoff KL, Warner ME, Posner KL, Stephens L, Domino KB. Pulmonary Aspiration of Gastric Contents: A Closed Claims Analysis. Anesthesiology. 2021 Aug 1;135(2):284-291. doi: 10.1097/ALN.0000000000003831. PMID 34019629
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530
- [Background] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Background] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Background] Bolondi L, Bortolotti M, Santi V, Calletti T, Gaiani S, Labo G. Measurement of gastric emptying time by real-time ultrasonography. Gastroenterology. 1985 Oct;89(4):752-9. doi: 10.1016/0016-5085(85)90569-4. PMID 3896910